CLINICAL TRIAL: NCT04923828
Title: Children's Hospital of Fudan University
Brief Title: Chinese PICU Collaborative Network on Pathogens and Drug Resistance of Severe Infections
Status: Recruiting | Type: Observational
Sponsor: Guoping Lu (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other); Ningbo Women & Children's Hospital (Other); Anhui Provincial Children's Hospital (Other); Xian Children's Hospital (Other Government); The Children's Hospital of Zhejiang University School of Medicine (Other); Qilu Children's Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Guoping Lu, Chief of PICU, Children's Hospital of Fudan University
Organization: Children's Hospital of Fudan University (Other)
Other Study IDs: fdpicu-21
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Severe Infection
Keywords: PICU; pathogen; severs infection; drug resistance
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate PICUs in major cities in China by establishing a high-quality standardized clinical database of PICU inpatients Incidence, fatality rate, pathogen distribution, anti-infective treatment of community-acquired/nosocomial infections in inpatients.

DETAILED DESCRIPTION:
All patients admitted to the PICU during January 1, 2016 to December 31 2025 were included in the study, and all patients were followed up until death or PICU withdrawal. To establish the standardized Access database collected patients' general information, infection, PICU treatment, catheter, and short-term Prognosis and other clinical data.

ELIGIBILITY:
Inclusion Criteria:

* PICU patients with severe infection

Exclusion Criteria:

* Non-infected patient

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PICU patients with severe infection
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathogenic spectrum of PICU severe infection | 2016-2025
  the 10 years of pathogenic spectrum of PICU severe infection

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China